CLINICAL TRIAL: NCT06593210
Title: Safety and Immunogenicity of Non-live, Adjuvanted Respiratory Syncytial Virus (RSV) Vaccine in Allogeneic Stem Cell Transplant and Lung Transplant Recipients
Brief Title: RSV Vaccine in Transplant Recipients
Acronym: RSVax
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The PSI Foundation, Ontario (Unknown); University of British Columbia (Other)
Responsible Party: Principal Investigator, Victoria Hall, Clinician-Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-5021
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Vaccine Response Impaired; Respiratory Syncytial Virus Infections; Immune Suppression
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Adjuvants, Pharmaceutic; arexvy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RSV vaccine group (Experimental): Single arm open label study of RSV vaccine to all adult transplant participants enrolling into the study.
  Interventions: Biological: Adjuvant, non-live RSV vaccine

INTERVENTIONS:
Biological: Adjuvant, non-live RSV vaccine — One dose of arexvy vaccine to transplant recipients.
  Other Names: Arexvy

SUMMARY:
Adjuvant, non-live RSV vaccine will be administered to adult lung and allogeneic hematopoietic stem cell transplant recipients. The safety and immunogenicity of this intervention will be studied. Blood work will be collected before and after the intervention, to assess humoral and cellular immunity. Participants will be followed for adverse reaction, hospitalization, RSV breakthrough infection, graft rejection or graft versus host disease. This study has Health Canada and UHN REB approval.

DETAILED DESCRIPTION:
This is a single-arm, open-label, investigational and interventional study to determine the immunogenicity of one dose of RSV vaccine in adult Allogeneic Stem Cell Transplant (alloSCT) or lung transplant (LT) recipients.Patients at least 18 years of age will receive a single dose of adjuvanted RSV vaccine (RSVPreF3, Arexvy, GSK). This vaccine is currently approved in Canada for adults over 60 years of age. Therefore, administration to adult transplant recipients between the age of 18 and 60 years of age is considered off-label. We have ethics approval to conduct this study from UHN and a No Objection Letter from Health Canada.

Study investigators (physicians) will perform the vaccination at hospital outpatient clinics.

Whole blood (total 30mL or 3 tubes) will be collected prior to vaccination and then at 4 weeks, 6 months and 12 months post-vaccination for humoral and cell-mediated immunity assessment. At each time point, 1 red-top blood tube (6mls) for serum and 2 green-top sodium heparin (9mls) blood tubes for plasma and peripheral blood mononuclear cells (PBMCs) will be collected.

Eligible patients will be screened as per the inclusion and exclusion criteria detailed in the screening log. After written informed consent and enrolment, the patient will be allocated a study code and data will be collected for demographics, including age, sex, gender identity, race, language spoken at home, immunosuppression at time of vaccination, time from transplant, immunosuppression regimen at time of transplant, underlying disease, recent lymphocyte count and immunoglobulin levels at the time of vaccination and follow up blood work. For alloSCT recipients, treatment history for Graft versus Host Disease (GvHD) and underlying disease status will be collected. For LT recipients, information regarding recent lung function and rejection episode(s) will be collected. Patients will be contacted at 6 weeks post-vaccination to determine the rates of adverse events including hospitalizations, cardiac, or neurologic events. Patients will then be contacted at 12 months and interviewed to determine whether they had a diagnosis of RSV infection following vaccination. Total follow-up time for each patient will be 1 year from vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Stable outpatient lung transplant recipients more than 3 months post-transplantation and stable outpatient allogeneic HCT recipients more than 6 months post-transplantation
* Adult equal or over 18 years of age
* Able to comply with blood work at 4-6 weeks post-vaccination
* Able to provide informed consent

Exclusion Criteria:

* Currently pregnant or planning to conceive or breastfeeding
* IVIg or plasmapharesis in last 30 days or expecting in next 30 days
* Previous rituximab in last 6 months
* Active CMV infection with VL > 1000 IU/ml
* Diagnosis of RSV in the past 90 days
* Unwell with acute infection (respiratory or other)
* Any vaccination in last 2 weeks
* History of severe allergic reaction (anaphylaxis) to any vaccination
* Active rejection in last 30 days for lung transplant recipient
* Active GvHD or poor graft function for alloSCT recipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Humoral immunogenicity | 4 weeks after dose 1
  Neutralizing antibody response

SECONDARY OUTCOMES:
Cellular immunogenicity | 4 weeks after dose 1
  T cell immune response
Safety of the vaccine | 7 days after dose 1
  Side effects after vaccine
Long-term safety | 1 year post dose 1
  Hospitalization, adverse events, RSV breakthrough infection, GvHD, graft rejection
Durability of immunity | 12 months
  Humoral and cellular immunogenicity at 6 and 12 months post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Victoria G Hall, MBBS, Principal Investigator — UHN Toronto
Locations (1):
- University Health Network, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No